CLINICAL TRIAL: NCT00689585
Title: A Single Centre. Parallel-Group, Double-Blinded, Randomized, Placebo-Controlled Pilot Clinical Trial on Ethosuximide for the Treatment of Complex Regional Pain Syndrome (CRPS)
Brief Title: Safety and Efficacy Study of Ethosuximide for the Treatment of Complex Regional Pain Syndrome (CRPS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficult and enrolment low: decision was made to stop the study.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other)
Responsible Party: Mark A. Ware, Prinicipal Investigator, McGill University Health Centre - Pain Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN#07-062
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Complex Regional Pain Syndrome; Reflex Sympathetic Dystrophy; RSD; Chronic Pain; Ethosuximide; Zarontin; Anticonvulsant
MeSH Terms: conditions — Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy; Chronic Pain | interventions — Ethosuximide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Ethosuximide

INTERVENTIONS:
Drug: Placebo — 250mg matching placebo capsules
  Arms: 1
Drug: Ethosuximide — 500-1500mg/day over a 1-5 week dose titration period until maximal tolerated dose (MTD) attained, followed by 1 week MTD plateau period.
  Other Names: Zarontin
  Arms: 2

SUMMARY:
Pain remains the most debilitating symptom for adult patients suffering from complex regional pain syndrome (CRPS). Most CRPS patients gain little to no relief from current painkillers. The purpose of this study is to evaluate the efficacy and safety of ethosuximide in search of much-needed adjunctive therapy to relieve the pain and suffering associated with CRPS.

DETAILED DESCRIPTION:
This is a single centre, parallel-group, double-blind, randomized, placebo-controlled pilot clinical trial for adults suffering from complex regional pain syndrome (CRPS).

Twelve (12) subjects diagnosed with CRPS will be enrolled and randomized to receive orally, either ethosuximide or placebo. If the maximum trial medication dosage (1500mg) is reached, the subject will be in the study for a maximum of 10 weeks from screening (Clinic Visit 1) to the end of the drug cessation period. The minimum period a subject could complete the study would be 4 weeks presuming they were not previously on any disallowed drugs and only found the 500mg dose tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 years old;
* Diagnosis of Complex Regional Pain Syndrome (CRPS) using International Association for the Study of Pain criteria >6 months;
* Normal liver function (AST level <3x normal level);
* Normal kidney function (serum creatinine <133µmol/L);
* Full blood count, haematocrit >38%;
* Willing and able to give informed consent and of completing study questionnaires;
* Stable (no change in past two months) but suboptimal pain pharmacotherapy (i.e. additional pain control felt by patient and physician to be necessary);
* Able to attend research centre according to the visit schedule;
* Women of child-bearing potential must be using a reliable form of contraception i.e. oral contraceptives, a barrier method (condom or diaphragm), intra-uterine device or abstinence.

Exclusion Criteria:

* Optimal response to opioids, antidepressants, anticonvulsants or anti- inflammatory medications;
* Any history or indication of kidney or liver disease;
* Any history of alcohol abuse;
* Presence of diabetes;
* Subjects taking other anti-epileptic drugs, including gabapentin, pregabalin, topiramate, phenytoin, carbamazepine, and oxcarbazepine;
* Pregnancy (a serum bHCG pregnancy test will be performed as part of the initial blood panel);
* Known or suspected allergy to succinimides, ethosuximide, methsuximide (Celontin®), phensuximide;
* Any history of mental illness or disorder, which in the investigators opinion, interferes with the subjects ability to accurately report treatment response;
* Participation in other clinical trial in the 30 days prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (500mg-1500mg per day) and Safety profile | up to 10 weeks
  Primary outcomes will consist of the dose attained during the study and the safety (adverse event) profile. Maximum timeframe on study drug is 6 weeks. Adverse events will be collected up to one month after the trial period ends.

SECONDARY OUTCOMES:
Pain Intensity Scores on the Visual Analogue Scale (VAS) | up to 7 weeks
  Pain Intensity captured on Day 1 (First study visit post-disallowed drug cessation period) and 7 days after maximal-tolerated dose attained (Final Study Visit)
Pain Intensity Scores on the Numerical Rating Scale (NRS) | up to 5 weeks
  Pain Intensity using the Numerical Rating Scale will be captured by telephone every week during dose titration period (Days 3 and 6).
Neuropathic Pain Symptom Inventory (NPSI) | up to 7 weeks
  Day 1 (First study visit post-disallowed drug cessation period) and 7 days after maximal-tolerated dose attained (Final Study Visit)
Short Form 12v2 (SF-12v2) | up to 7 weeks
  Quality of Life measured on Day 1 (First study visit post-disallowed drug cessation period) and 7 days after maximal-tolerated dose attained (Final Study Visit)
Short Form McGill Pain Questionnaire (SF-MPQ) | up to 7 weeks
  Day 1 (First study visit post-disallowed drug cessation period) and 7 days after maximal-tolerated dose attained (Final Study Visit)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Ware, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada